CLINICAL TRIAL: NCT01070368
Title: Accuracy Of Skin Prick Test Using In-house Wheat Extract For The Diagnosis Of IgE-mediated Wheat Allergy: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, nittida pannakapitak, Principal investigator, Mahidol University
Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 231/2552(EC4)
Record Dates: First submitted 2010-02-16; First posted 2010-02-18 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Wheat Allergy
Keywords: skin test; open wheat challenge
MeSH Terms: conditions — Wheat Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Food challenge, skin test (Experimental): Skin test by two extract commercial, and in-house extract. and open challenge with wheat (except in patient with history of wheat anaphylaxis: assume as challenge positive)
  Interventions: Other: Commercial extract and in-house wheat extract

INTERVENTIONS:
Other: Commercial extract and in-house wheat extract — Patients with a history of wheat allergy underwent two skin test extracts, and open challenge with wheat. A blood test for specific IgE was performed in the same time.

SUMMARY:
Nowadays, commercial wheat extract is widely accessible, and is used for skin prick test for wheat allergy. However, commercial wheat extracted for skin prick test have less precise test result compared to extract from omega-5 gliadin, which is one of the major allergen with immediate wheat allergy.

ELIGIBILITY:
Inclusion Criteria:

* A patient with the age of 1-15 year old
* A history of symptoms that suspected of type 1 hypersensitivity (eg. Urticaria, angioedema, wheezing, anaphylaxis) occur within 4 hours after wheat ingestion.
* Patients attend in allergy clinic, pediatric department, Siriraj hospital since 2007-2012

Exclusion Criteria:

* First sign and symptom happens more than 4 hours since wheat ingestion
* Have underlying disease such as heart disease, epilepsy etc.
* Have contraindication for performed skin prick test

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2009-06; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
correlation skin test result and food challenge result | 3 year

SECONDARY OUTCOMES:
comparison of skin test result and specific IgE to challenge result | 3 year

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric department, Faculty of medicine Siriraj hospital, Mahidol university, Bangkok, Thailand